CLINICAL TRIAL: NCT04437147
Title: The Effect of Probiotics on Functional Constipation in Adults: Double-blind, Randomized, Placebo-controlled Study
Brief Title: Effect of Probiotics on Functional Constipation in Adults
Acronym: PROBCON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Luciane Cruz Lopes (Other)
Responsible Party: Sponsor-Investigator, Luciane Cruz Lopes, Principal Investigator: Fabiana Cristina Rosa Mitelmão, University of Sorocaba
Organization: University of Sorocaba (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Fabiana Rosa
Record Dates: First submitted 2020-06-03; First posted 2020-06-18 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Functional Constipation
Keywords: Lactobacillus; Bifidobacterium

STUDY DESIGN:
Intervention Model Description: Interventions: in particular, subjects were divided into 3 groups: i) 50 subjects in the group A will receive placebo, ii) 50 subjetcs in the group B will receive mixed L. acidophilus LA 02 ID 1688, B. bifidum BB 01 ID 1722 and L. rhamnosus LR 04 ID 1132 (1 x 10⁹ colony-forming units/d of each strain) and 50 subjects em the group C will receive L. acidophilus LA 02 ID 1688, B. bifidum BB 01 ID 1722, L. rhamnosus LR 04 ID 1132, L. paracasei LPC 00 ID 1076, B. longum BL 03 ID 1152, B. lactis BS 01 ID 1195, L. casei LC 03 ID 1872, B. animalis LMG 10508 (1 x 10⁹ colony-forming units/d of each strain) for 30 days. At the beginning of the interventional study, the healthy status of volunteers will be evaluated by a complete, laboratory and by the clinical evaluation by the doctor using as reference ROMA IV for intestinal constipation. Exclusion criteria will be items of gastrointestinal diseases, pregnant and antibiotic intake.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The phisician (care provider), the research subjects (participants) and outcome assessor (had access to the results) will be blinded. All groups received sachets with the same characteristics (taste and packaging) different only in the numbering of the manufacturing batches. The phisician separated each volunteer in according to lot number corresponding to the randomisation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): a) Control placebo (P1) Component Vitamin C (Ascorbic acid) 45 mg,Vitamin B1 (Thiamine) 1.1 mg, Vitamin B2 (Riboflavin) 1.1 mg,Vitamin D-3 40,000,000 IU / GR (Cholecalciferol) 34 mcg, Magnesium hydroxide 0.3 g, Calcium Carbonate 0.5 g, Natural Vanilla Flavor Powder 0.03 g,Fos (Fructooligosaccharides) qsp 3 g, for 30 days, once a day by sachet
  Interventions: Dietary Supplement: Placebo
- 3 Billion CFU strains of probiotics (Active Comparator): b) 3 Billion CFU (P2) Component Lactobacillus acidophilus LA 02 ID 1688 1 billion CFU,Bifidobacterium bifidum BB 01 ID 1722 1 billion CFU, Lactobacillus rhamnosus LR 04 ID 1132 1 billion CFU,Vitamin C (Ascorbic acid) 45 mg,Vitamin B1 (Thiamine) 1.1 mg, Vitamin B2 (Riboflavin) 1.1 mg,Vitamin D-3 40,000,000 IU / GR (Cholecalciferol) 34 mcg, Magnesium hydroxide 0.3 g, Calcium Carbonate 0.5 g, Natural Vanilla Flavor Powder 0.03 g,Fos (Fructooligosaccharides) qsp 3 g, for 30 days, once a day by sachet
  Interventions: Dietary Supplement: 3 Billion UFC strains of probiotics
- 8 Billion CFU strains of probiotics (Active Comparator): c) 8 Billion UFC (P3) Component Lactobacillus paracasei LPC 00 ID 1076 1 billion CFU;Bifidobacterium longum BL 03 ID 1152 1 billion CFU; Bifidobacterium lactis BS 01 ID 1195 1 billion CFU;Lactobacillus casei LC 03 ID 1872 1 billion CFU; Bifidobacterium animalis LMG 10508 1 billion CFU; Lactobacillus acidophilus LA 02 ID 1688 1 billion CFU,Bifidobacterium bifidum BB 01 ID 1722 1 billion CFU, Lactobacillus rhamnosus LR 04 ID 1132 1 billion CFU,Vitamin C (Ascorbic acid) 45 mg,Vitamin B1 (Thiamine) 1.1 mg, Vitamin B2 (Riboflavin) 1.1 mg,Vitamin D-3 40,000,000 IU / GR (Cholecalciferol) 34 mcg, Magnesium hydroxide 0.3 g, Calcium Carbonate 0.5 g, Natural Vanilla Flavor Powder 0.03 g,Fos (Fructooligosaccharides) qsp 3 g, for 30 days, once a day by sachet
  Interventions: Dietary Supplement: 8 Billion UFC strains of probiotics

INTERVENTIONS:
Dietary Supplement: Placebo — Fibers with vitamins and minerals will be administered for 30 days once a day in sachets
  Other Names: Group Placebo
  Arms: Placebo
Dietary Supplement: 3 Billion UFC strains of probiotics — Fibers with vitamins and minerals will be administered for 30 days once a day in sachets with 3 billion CFU strains of probiotics
  Arms: 3 Billion CFU strains of probiotics
Dietary Supplement: 8 Billion UFC strains of probiotics — Fibers with vitamins and minerals will be administered for 30 days once a day in sachets with 8 billion CFU strains of probiotics
  Arms: 8 Billion CFU strains of probiotics

SUMMARY:
Introduction:

Functional constipation is a symptom-based gastrointestinal disorder without an organic origin (eg, bowel obstruction). It has a prevalence of 14% in adults.

Objective:

The objective of trial is to evaluate the efficacy and safety of two different probiotic blends in adults subjects with functional constipation.

Methods:

A double-blind, randomized, placebo-controlled study will be conducted for up to two years to evaluate the efficacy of two different probiotic mixtures: (Mixture 1) Lactobacillus acidophilus, Bifidobacterium bifidum and Lactobacillus rhamnosus (3 billion CFU); (Mixture 2) Lactobacillus acidophilus, Bifidobacterium bifidum, Lactobacillus rhamnosus, Lactobacillus paracasei, Bifidobacterium longum, Bifidobacterium lactis, Lactobacillus defensis, Bifidobacterium animallis (8 billion CFU).

DETAILED DESCRIPTION:
The study involve 150 healthy volunteers with functional constipation.The sample size was based on literature reviews of the probiotics' effect comparing the differences between means.

After confirmation of eligibility and obtaining written informed consent, the patients will be randomized (stratification for blocks) to recivied the interventions. The patients and the phisician will be blinded to the treatment received. The eligible patients will be allocated (1:1:1) to treatment with either the probiotics supplements or placebo. Subjects will be instructed to ingest one sachet before breakfast, by mixing the powder in water and drinking it. The sachets will be stored at room temperature.

Data handling and record keeping Case report forms will be used to record data for all participants, and will be completed by the research doctor, who will also enter the data into an electronic database.

Study schedule and location After inclusion, all further treatments will be managed at the primary care center where the subject was recruited. A research doctor and a research pharmacist will be responsible for all contacts with patients.

Local of study development Recruitment of patients to this study will be made by collaboration with the Gastroenterolgy Clinic at Avenue Dr Armando Sales de Oliveira 371, Trujilo, Sorocaba, State of São Paulo, Brazil from March 2020 to April 2020. Sorocaba is a Brazilian municipality in the interior of the state of São Paulo. It is the fourth most populous in the interior of São Paulo in the Southeast of the country, and the most populous in the southern region of São Paulo, with a population of 671,186 inhabitants, estimated by IBGE for July 1, 2018.

For comparison of three groups, an independent t-test will be applied for continuous variables and Mann-Whitney for non-continuous variables. Analysis of adverse events (if any) will be performed using Chi-Square test and Fisher's exact test following assumptions of randomness, independence and size. Significance differences will be set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

-Clinical diagnosis of functional constipation according to Rome IV. Granting of written informed consent.

Exclusion Criteria:

* Presence of gastrointestinal diseases
* Ingestion of antibiotics or dietary supplements containing probiotics or prebiotics in the last 15 days
* Pregnancy.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-01-28 (Actual)

PRIMARY OUTCOMES:
Changed in the number of Bowel movements. Changed for more than 3 per week was considered a clinical response. | 30 days
  Changed number of bowel movements evaluated weekly
Change in the Bristol stool form scale at 4 weeks after Probiotics. Recovery to types 3-4 was considered a clinical response. | 30 days
  The Bristol scale ranges from 1-7, with 1-2 being constipated, 3-5 normal and 6-7 diarrhea.

SECONDARY OUTCOMES:
Subject withdrawal | 30 days
  The volunteers can withdraw from the study at any time by their own request, or can be withdrawn at any time at the discretion of the investigator for safety. Volunteers will also be withdrawn from the study in the event of treatment interruption for any reason, whether due to forgetfulness or to experiencing undue intestinal discomfort
Adverse events | 30 days
  Adverse events are undesirable signs or symptoms that occur during the study and whose cause may or may not be causal related to the treatment. All adverse events considered possibly, probably or related to the test product will be noted down on the patient's form.
Serious adverse events | 30 days
  Serious adverse events are defined as events that are fatal, life-threatening, disabling or result in hospitalization or prolonged stay, or result in malformation, whether related to the test product or otherwise.
  According to previous studies, probiotics are safe and any serious adverse event that could possibly, probably or be related to the test products will be considered unexpected. All unexpected serious adverse events will be reported to the physician. Any serious adverse event that may be related to the test product will immediately lead to discontinuation of the test product

CONTACTS AND LOCATIONS:
Overall Officials: Fabiana R MITELMAO, master, Principal Investigator — UNIVERSIDADE DE SOROCABA
Locations (1):
- Universidade de Sorocaba, Sorocaba, São Paulo, Brazil

REFERENCES:
- [Derived] Mitelmao FCR, Hackel K, Bergamaschi CC, Gerenutti M, Silva MT, Balcao VM, Vila MMDC. The effect of probiotics on functional constipation in adults: A randomized, double-blind controlled trial. Medicine (Baltimore). 2022 Oct 28;101(43):e31185. doi: 10.1097/MD.0000000000031185. PMID 36316826